CLINICAL TRIAL: NCT02681887
Title: Effect of Melatonin on Cardiometabolic Risk- FULL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, John P. Forman, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2015P002524
Record Dates: First submitted 2016-02-03; First posted 2016-02-15 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Obesity; Prediabetic State
MeSH Terms: conditions — Obesity; Prediabetic State | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo tablet identical to Circadin by mouth each day before bedtime for 12 weeks
  Interventions: Drug: Placebo
- Melatonin (Experimental): Circadin, controlled release melatonin tablet 2mg by mouth each day before bedtime for 12 weeks
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin — Circadin, controlled release melatonin tablet 2mg by mouth each day before bedtime for 12 weeks
  Other Names: Circadian
  Arms: Melatonin
Drug: Placebo — placebo tablet identical to circadian
  Arms: Placebo

SUMMARY:
In a 12 week double-blind, placebo-controlled randomized trial, 120 subjects with obesity (BMI≥30 kg/m2) and pre-diabetes (HbA1c, 5.7-6.4%) will be randomly assigned 1:1 to receive either placebo or 2 mg of controlled-release melatonin, taken orally every evening 1 hour before bed. The investigators will assess melatonin's effect on insulin sensitivity by performing a hyperinsulinemic euglycemic glucose clamp and β-islet cell function measured using a hyperglycemic clamp, as a primary endpoint. The investigator will also evaluating melatonin supplementation's effect on mean 24-hour ambulatory blood pressure, nocturnal blood pressure, and potential intermediates including endothelial function using brachial ultrasound, catecholamine production using 24-hour epinephrine and norepinephrine excretion, and renin-angiotensin system activation using measurements of plasma renin activity, angiotensin II, and urine aldosterone excretion. The final endpoint will be to evaluate melatonin supplementation's effect on cellular cytokine and CC family chemokine expression as well as high sensitivity C-reactive protein, IL-6, and TNF-α.

There will be a 24 week cohort phase as an extension of the trial. This will be an open-label prospective study of 50 subjects recruited from the trial who will take 2 mg of controlled-release melatonin nightly for 24 weeks after completion of the 12-week trial. At the end of the cohort-phase (36 weeks after entry in the trial), the investigators will again assess the extended use of melatonin supplementation on 24-hour BP, and glycemic control (HbA1, fasting glucose).

DETAILED DESCRIPTION:
All participants will be recruited locally in the Boston area, and all study visits and procedures will be conducted through Partners and the Harvard Catalyst.

Briefly, the trial-phase will consist of four visits, two as outpatient, and two as inpatient. The cohort-phase will consist of two additional outpatient visits. The screening outpatient visit will involve history taking, physical examinations (when appropriate), phlebotomy to measure circulating factors and urine pregnancy testing for female subjects. The 6-week outpatient check-up visit will be with a study coordinator. In addition to evaluating for adverse effects, the coordinator will perform a pill-count. Phlebotomy will be performed to measure circulating factors. The two inpatient visits will require two overnight stays each; the procedures performed for these two inpatient stays will be identical, and will include: timed urine collection, measurement of brachial artery flow mediated dilation, phlebotomy (including an IV protocol using low dose heparin), hyperinsulinemic euglycemic clamp, hyperglycemic clamp, central blood pressure, and placement of an ambulatory blood pressure monitor that the participant will wear home for 24 hours and return by pre-paid FedEx mailer. We will take blood samples at each visit, collecting about 54 tablespoons (798.5 mL) of blood over the 36-week course of the study.

Outpatient visits: A screening visit will be scheduled when a participant expresses interest in the study and is deemed potentially eligible by the study coordinator after a telephone interview. At the screening visit, a study physician will obtain informed consent. Thereafter, a study physician will conduct a history and physical examination, and phlebotomy will be performed. Female subjects will provide urine for pregnancy testing. The purpose of the screening visit is to evaluate potential volunteers based upon the inclusion and exclusion criteria listed above, and to explain the purpose and procedures of the study to the volunteers. If someone is eligible and willing, a baseline inpatient visit will be scheduled.

A 6-week check up will be scheduled after the subject completes the initial inpatient visit. In addition to evaluating for adverse effects, the coordinator will perform a pill-count. Phlebotomy will be performed to measure circulating factors.

For the cohort phase, 24- and 36-week check up visits will be scheduled after the subject completes the final inpatient visit. At these visits, in addition to evaluating for adverse effects, the coordinator will perform a pill-count. Phlebotomy will be performed to measure circulating factors.

Inpatient visits: Prior to each inpatient visit, participants will be mailed 9 bouillon packets (containing 50 mmol of sodium each) and instructed to consume 3 packets each day for three days prior to admission to the Clinical Trials Center; the purpose of this is to achieve high sodium balance, which is necessary for our measurements of the renin-angiotensin system. The high sodium diet will be continued during the inpatient setting. Female subjects will have a urine pregnancy test done at admission. The following measurements will be performed during the two inpatient visits, and the changes in these measurements (comparing the baseline value with the 8-week value) are the endpoints for this study:

1. A hyperinsulinemic euglycemic clamp will be performed to measure peripheral insulin sensitivity. Intravenous catheters are placed within each arm (one for infusion, and one for blood collection). Then, a compound called insulin (supplied by the Investigational Drug Service (IDS)) is infused as a loading dose followed by a continuous infusion to achieve a steady state condition. Blood samples are collected every 5 minutes, and glucose levels are measured. Blood glucose levels will be controlled by the infusion of a 20% dextrose solution. The mean dextrose infusion rate (M) over the period between 120 and 180 minutes will be used to measure insulin sensitivity. At 180 minutes, the study will conclude, and both infusions will be stopped.
2. A hyperglycemic clamp will be performed to measure pancreatic β-cell function. Intravenous catheters are placed within each arm (one for infusion, and one for blood collection). After a baseline period of 30 minutes, the blood glucose level is increased with a loading dose of dextrose followed by a continuous infusion to achieve a steady state condition. Blood samples are collected every 5 minutes, and glucose levels are measured. Insulin levels are measured at 0, 2.5, 5.0, 7.5, 10, 20, 40, 60, 80, 100, 120, 140, 160, 180 minutes after the infusion. The 1st-phase insulin release is the sum of the plasma insulin concentrations at 2.5, 5.0, 7.5 and 10 minutes. The 2nd-phase is the average plasma insulin concentration during the final hour.
3. Endothelial-dependent vasodilation using brachial artery diameter will be measured by ultrasound. A blood pressure cuff will be inflated on the arm to a supra-systolic pressure for 5 minutes. This results in vasodilation of the downstream blood vessels. Following release of the cuff, there is usually a 6 to 10-fold increase in flow through the brachial artery, i.e., reactive hyperemia. Flow is a physiologic stimulus that releases nitric oxide and causes dilation of the brachial artery, and hence, an increase in the diameter of the brachial artery; this can be measured using ultrasound. The maximal increase in brachial artery diameter occurs at one minute of reactive hyperemia and this dilation is mediated by nitric oxide. Endothelium-independent vasodilation (as a positive control) will be assessed by measuring brachial artery diameter under basal conditions and 3 minutes following the administration of sublingual nitroglycerin (0.4 mg). Maximal brachial artery dilation occurs 3 to 4 minutes after the administration of sublingual nitroglycerin.
4. Central aortic blood pressure measurement: The SphygmoCor XCEL System is a portable machine that will be used to measure central aortic blood pressure at each of the inpatient visits (this machine is FDA approved for measurement of central blood pressure). A thin pillow is placed under the subject's arm to align the arm with the heart. A blood pressure cuff is placed on the patient's arm, over the brachial artery to obtain this measurement. The entire procedure will take approximately 10 minutes to perform. Coded data is automatically stored via the SphygmoCor XCEL System and can be downloaded onto a secure research computer for storage and analysis.
5. Phlebotomy will be performed to measure circulating melatonin, plasma renin activity, and angiotensin II. These assays are markers of the systemic renin angiotensin system. Phlebotomy will also measure adiponectin, leptin, ghrelin, and HbA1c. These assays are markers of glucose homeostasis and insulin sensitivity. In addition, intravenous access will be placed to permit blood draws every 2 hours from 7 pm until 9 am the following morning (ie, the morning of day 1). These nocturnal blood draws will be used to measure nocturnal serum melatonin levels. In order for these blood draws to be completed without entering the subject's room and possibly waking the subject, a specialized circadian IV protocol will be used whereby an antecubital IV line will be secured with a kerlix wrap and connected to a 12 foot IV tubing that will traverse a metal window in the wall that was constructed especially for such purposes and that is present in patient rooms in the BWH CCI. Patency of the IV tubing during the night will be ensured by infusing a low dose of unfractionated heparin (approximately 200 units per hour). The heparin will be stopped and the IV converted to a standard IV at approximately 9 am on Day 1. This is standard protocol in the BWH CCI for measuring overnight melatonin concentrations.
6. A 24-urine will be collected to measure excretion of epinephrine, norepinephrine, and aldosterone.
7. Ambulatory blood pressure (for 24 hours) will be measured using a standard technique employed commonly in clinical practice. An ambulatory blood pressure monitor will be placed on the participant's arm before the participant is discharged from the inpatient visit; the participant will also be instructed on its appropriate use, including how to shut the monitor off after a 24-hour period. The participant will be discharged from the inpatient visit with the cuff in place and will be given a pre-paid FedEx mailer so that the monitor can be returned to the study coordinator for data download and re-use.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* body mass index (BMI) >30
* HbA1c 5.4-6.4%
* if hypertensive, BP <150/90

Exclusion Criteria:

* Use of a melatonin supplement
* Current use of anticoagulants
* Use of hypoglycemic or antihypertensive meds
* Current or prior history of diabetes mellitus, or random serum glucose ≥ 200 mg/dL
* Major bleeding event in the past 60 days
* Recent (past 2 weeks) or upcoming travel across time zones
* Known obstructive sleep apnea or use of continuous positive airway pressure
* Known heparin allergy
* Hepatic impairment
* Estimated GFR <60 mL/min/1.73m2
* Pregnant
* Job requires rotating night shifts
* Preexisting lung disease requiring oxygen
* Active chronic or acute infection
* Preexisting CVD
* Known melatonin allergy
* Bariatric surgery within the prior 12 months
* Preexisting hemoglobinopathy
* Use of weekly or daily NSAID for chronic pain
* Use of cholesterol lowering medications
* Active or uncontrolled psychotic disorder
* Use of hypnotic medications
* Active or uncontrolled bipolar illness
* Active or uncontrolled depression
* Recent (within the past three months) blood donation or plan to donate blood during study period
* Use of a phosphodiesterase inhibitor
* Active malignancy within the prior 5 years
* Hypertension (>150/90)
* Currently lactating (women)
* History of stroke
* Hematocrit <36 (women) or <41 (men)
* Thrombocytopenia or other bleeding disorders
* Surgery in the past 60 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
change in insulin sensitivity | 12 weeks
  measure insulin sensitivity using hyperinsulinemic clamp
change in beta-islet cell function | 12 weeks
  measure beta-iset cell function measured using a hyperglycemic clamp

SECONDARY OUTCOMES:
change in 24 hour ambulatory blood pressure | 12 weeks
  evaluate the effect of supplementation on 24-hour ambulatory blood pressure
change in nocturnal blood pressure | 12 weeks
  evaluate the effect of supplementation nocturnal blood pressure
change in endothelial dependent vasodilation | 12 weeks
  Measurements of the brachial diameter will be made under basal conditions and during reactive hyperemia following five minutes of ischemic stimulus
change in endothelial independent vasodilation | 12 weeks
  measuring brachial artery diameter under basal conditions and 3 minutes following the administration of sublingual nitroglycerine (0.4mg)
change in catecholamine production | 12 weeks
  using 24 hour urine collection, measure catecholamines from (epinephrine, norepinephrine and dopamine) using a RIA
change in plasma renin level | 12 weeks
  effect of melatonin on RAS
change in angiotensin II level | 12 weeks
  effect of melatonin on RAS
change in cellular cytokine level | 12 weeks
  effect of melatonin on inflammatory markers
change in CC family chemokine expression | 12 weeks
  effect of melatonin on inflammatory markers
change in high sensitivity CRP | 12 weeks
  effect of melatonin on inflammatory markers
change in IL-6 level | 12 weeks
  effect of melatonin on inflammatory markers
change in TNF-alpha | 12 weeks
  effect of melatonin on inflammatory markers

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States